CLINICAL TRIAL: NCT02900612
Title: Effects of Two Aquatic Training Models in Physiological Parameters of Elderly Dyslipidemic Women: a Randomized Controlled Clinical Trial.
Brief Title: Effects of Two Aquatic Training Models in Physiological Parameters of Elderly Dyslipidemic Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0547
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Dyslipidemias
Keywords: dyslipidemias,; aging; water aerobics training; resistance aquatic training; lipid profile
MeSH Terms: conditions — Dyslipidemias | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- WA (Water Aerobics Training) (Experimental): Water aerobics training.
  Interventions: Other: Water aerobics training.
- WR (Water Resistance Training) (Experimental): Resistance aquatic training.
  Interventions: Other: Water resistance training.
- CG (Control Group) (Active Comparator): Control Group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Water aerobics training. — The WA group will be trained adopting the interval method, performing six blocks of five minutes each one, alternating four minutes at intensities corresponding to 90 to 100% of the heart rate corresponding to the second ventilatory threshold (HRVT2) and one minute at intensities between 80 and 90% HRVT2.
  Other Names: WA
  Arms: WA (Water Aerobics Training)
Other: Water resistance training. — The WR group will perform four to eight sets of 20 to 10 seconds along the macrocycle, always at maximal speed execution of the exercises.
  Other Names: WR
  Arms: WR (Water Resistance Training)
Other: Control Group — The control group will perform relaxation classes, including meditation, balance exercises, coordination exercises.
  Other Names: CG
  Arms: CG (Control Group)

SUMMARY:
This study aims to compare the effects of two water-based training models in physiological parameters of dyslipidemic elderly women. Thus, a randomized controlled clinical trial will be conducted in parallel with the participation of 45 dyslipidemic elderly women.

DETAILED DESCRIPTION:
The women will be randomly divided into three groups: water aerobics training (WA), resistance aquatic training (WR) and the third is the control group (who will perform relaxation sessions under water). The three groups will attend classes during 10 weeks, with two weekly sessions of 45 minutes each. The WA and WR groups will use the same four exercises in their training.

The WA group will be trained using the interval method, performing six blocks of five minutes each one, alternating four minutes at intensities corresponding to 90 to 100% of the heart rate corresponding to the second ventilatory threshold (HRVT2) and one minute at intensities between 80 and 90% HRVT2.

The WR group will perform four to eight sets of 20 to 10 seconds along the macrocycle, always at maximal speed execution of the exercises.

Will be measured, before and after the period of 10 weeks of intervention, biochemical, cardiorespiratory, neuromuscular and hemodynamic variables, parameters of quality of life and depressive symptoms in addition to the cardiovascular risk score of the participants of the three groups.

Data will be described by means values and lower and upper limits, with a 95% confidence interval. Comparisons between and within groups were performed using the method of generalized estimates of equations (GEE), with Bonferroni post hoc, adopting a 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* being female, aged between 60 and 75, sedentary (not practicing any kind of regular, supervised physical activity in the last three months), have any type of dyslipidemia.

Exclusion Criteria:

* women who are smokers, suffering from cardiovascular disease with associated complications and those with orthopedic diseases that prevented the practice of systematic physical exercise, users of hormone therapy drugs and lipid-lowering medications.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol (TC) Change | Change from baseline total cholesterol at 10 weeks
  This variable will be measured through blood collection after 12 hours fasting. The analysis will be performed through the enzymatic method using kits Siemens, in automated equipment Advia 1800.

SECONDARY OUTCOMES:
Triglycerides (TG) Change | Change from baseline triglycerides at 10 weeks
  This variable will be measured through blood collection after 12 hours fasting. The analysis will be performed through the enzymatic method using kits Siemens, in automated equipment Advia 1800.
High Density Lipoprotein (HDL) Change | Change from baseline HDL at 10 weeks
  This variable will be measured through blood collection after 12 hours fasting. The analysis will be performed through the enzymatic method using kits Siemens, in automated equipment Advia 1800.
C-Reactive Protein (CRP) Change | Change from baseline C-reactive protein at 10 weeks
  This variable will be measured through blood collection after 12 hours fasting. The analysis will be performed through the turbidimetric method in Cobas Mira Plus equipment, with the Biotechnical Kit for ultrasensitive C-reactive protein.
Low Density Lipoprotein (LDL) Change | Change from baseline LDL at 10 weeks
  This variable will be estimated by Friedewald equation.
Total Cholesterol/High Density Lipoprotein Ratio (TC/HDL ratio) Change | Change from baseline TC/HDL at 10 weeks
  This variable will be estimated by the simple division of variables.
Peak Oxygen Consumption (VO2peak) Change | Change from baseline VO2peak at 10 weeks
  This outcome will be measure through maximal progressive treadmill test, using the portable gas analyser VO2000 equipment.
Oxygen Consumption at anaerobic threshold (VO2VT2) Change | Change from baseline VO2VT2 at 10 weeks
  This outcome will be measure through maximal progressive treadmill test, using the portable gas analyser VO2000 equipment.
Heart Rate at anaerobic threshold (HRVT2) Change | Change from baseline HRVT2 at 10 weeks
  This outcome will be measure through maximal progressive treadmill test, using a heart rate monitor (POLAR, FT1).
Rest Heart Rate (HRrest) Change | Change from baseline HRrest at 10 weeks
  This outcome will be measure using a heart rate monitor (POLAR, FT1). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the heart rate.
Lipoprotein Lipase (LPL) Change | Change from baseline LPL at 10 weeks
  This variable will be measured through blood collection after 12 hours fasting. The analysis will be performed using the LPL ELISA kit (Cell Biolabs). The results will be read in a microplate reader (ELISA).
Maximal dynamic muscle strength of knees extensors (MSKE) Change | Change from baseline MSKE at 10 weeks
  This outcome will be measured through the one-repetition maximal test (1RM).
Maximal dynamic muscle strength of knees flexors (MSKF) Change | Change from baseline MSKF at 10 weeks
  This outcome will be measured through the one-repetition maximal test (1RM).
Maximal dynamic muscle strength of horizontal shoulder flexors (MSHSF) Change | Change from baseline MSHSF at 10 weeks
  This outcome will be measured through the one-repetition maximal test (1RM).
Rest Cardiac Output (COrest) Change | Change from baseline COrest at 10 weeks
  This outcome will be measured through Impedance Cardiography (Physioflow Lab-1 equipment). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the cardiac output.
Rest Stroke Volume (SVrest) Change | Change from baseline SVrest at 10 weeks
  This outcome will be measured through Impedance Cardiography (Physioflow Lab-1 equipment). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the stroke volume.
Peak Cardiac Output (COpeak) Change | Change from baseline COpeak at 10 weeks
  This outcome will be measured through Impedance Cardiography (Physioflow Lab-1 equipment), during a maximal progressive treadmill test.
Peak Stroke Volume (SVpeak) Change | Change from baseline SVpeak at 10 weeks
  This outcome will be measured through Impedance Cardiography (Physioflow Lab-1 equipment), during a maximal progressive treadmill test.
Rest Arterial Systolic Blood Pressure (SBPrest) Change | Change from baseline SBPrest at 10 weeks
  This outcome will be measured through blood pressure ambulatory monitor (Meditech, ABPM-04). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the arterial systolic blood pressure.
Rest Arterial Diastolic Blood Pressure (DBPrest) Change | Change from baseline DBPrest at 10 weeks
  This outcome will be measured through blood pressure ambulatory monitor (Meditech, ABPM-04). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the arterial diastolic blood pressure.
Cardiovascular Risk Score (CRS) Change | Change from baseline cardiovascular risk score at 10 weeks
  The Reynolds Risk Score Instrument will be used to estimate the cardiovascular risk.
Quality of Life Change | Change from baseline quality of life at 10 weeks
  The quality of life will be estimated using the Whoqol-Bref instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided